CLINICAL TRIAL: NCT01455155
Title: Efficacy of Creative Therapy for Stroke Patients
Brief Title: Creative Therapy to Affect Stroke Outcomes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si290/2011
Record Dates: First submitted 2011-10-15; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Stroke
Keywords: stroke; Art therapy; Music therapy; Creative therapy; Efficacy
MeSH Terms: conditions — Stroke | interventions — Reproductive Techniques, Assisted; Music Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Creative therapy (Experimental): Conventional physical therapy program (5 times/week) plus creative therapy (Art and Music) 2 times/week for 4 weeks
  Interventions: Other: Creative therapy (art and music therapy)
- Control (Active Comparator): Conventional physical therapy (5 times/week) for 4 weeks
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Creative therapy (art and music therapy) — Creative therapy composed of groups of activities relating to music and art sciences 8 sessions (2 sessions per week for 4 weeks) These activities emphasized on stimulating of cognition, physical, emotion, communication, social relationship, and spiritual domains.
  Arms: Creative therapy
Other: Physical therapy — Physical therapy composed of a series of physical therapy program including types of exercises and gait training if possible (5 times/week).
  Arms: Control

SUMMARY:
Stroke is one of the common diseases in the elderly. It is the third ranking cause of death and affects health care system in our country. The focal brain lesions encountered in patients with stroke can result in impairments in motor function, language, cognition, sensory processing, cognition and emotional disturbances. All of these conditions affect performance of functional activities. The abrupt change in the life situation of the stroke survivor impacts all phases of care. This may reduce a patient's quality of life.

Many innovative therapy techniques have been developed to help the restoration of lost functions and to aid in prevention and treatment of depression. Music and art therapy has been used in rehabilitation settings to stimulate brain functions involved in movement, cognition, speech, emotions, and sensory perceptions. However many research studies on the use of music and art therapy in rehabilitation of acquired brain injury have suffered from small sample size, making it difficult to achieve statistically significant results. In addition, differences in factors such as study designs, methods of interventions, and intensity of treatment have led to varying results.

DETAILED DESCRIPTION:
Our study focuses on the use of creative therapy with a patient diagnosed with stroke. Creative therapy refers to a group of techniques include art therapy, writing, movement therapy, role play, and music therapy that are expressive and creative in nature. The aim of creative therapies is to help patients find a form of expression beyond words or traditional therapy, such as cognitive or psychotherapy. These therapies use arts modalities and creative processes during intentional intervention in therapeutic, rehabilitative, community, or educational settings to foster health, communication, and expression.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients
* Duration of stroke >=1 month
* Age >=50 years
* Ability to follow command and communicable

Exclusion Criteria:

* Unstable medical conditions, including fever, uncontrolled hypertension
* Serious contact diseases, for example AIDS, TB
* Severe dementia or uncontrolled psychiatric problems

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-10 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Abbreviated Mental Score test (AMS) | 4 weeks
  The creative therapy will be considered success if the AMS increases after 4-week of treatment.

SECONDARY OUTCOMES:
Barthel index (BI) | 4 weeks
  The creative therapy will be considered success if the BI score increases after 4-week of treatment.
Hospital anxiety depression score (HADS) | 4 weeks
  The creative therapy will be considered success if the HADS decreases after 4-week of treatment.
Pictorial Thai Quality of Life score | 4 weeks
  The creative therapy will be considered success if the pictorial Thai Quality of Life score increases after 4-week of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Vilai Kuptniratsaikul, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand